CLINICAL TRIAL: NCT06733272
Title: The Relationship Between Healthy Lifestyle Behaviors, Physical Activity and Blood Tests in Pregnancy
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Collaborators: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Betul Ergun, Lecturer, Inonu University
Other Study IDs: Pregnancy
Record Dates: First submitted 2024-11-27; First posted 2024-12-13 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2024-11

CONDITIONS: Pregnancy
Keywords: Pregnancy; Blood Tests; Physical Activity; Healthy Lifestyle Behaviors
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Pregnancy is a significant phase in women's lives, marked by psychological, biological, and emotional changes. It lasts for approximately nine months and is divided into three trimesters. Identifying risk factors such as maternal age, gestational age, ethnicity, and lifestyle habits is crucial for managing pregnancy effectively. Anxiety, depression, and stress can significantly impact pregnancy-related responsibilities and overall well-being, making collaboration with a multidisciplinary healthcare team essential.

Physical activity during pregnancy offers numerous benefits, including better physical fitness, improved psychological health, weight management, and reduced risk of gestational diabetes. However, studies show that many women are not sufficiently active, particularly in the first trimester, where activity levels tend to be lower. Regular monitoring of thyroid function (TSH levels) and liver enzymes (ALT, AST) is essential to avoid complications, as pregnancy can affect thyroid function and liver health. Additionally, monitoring hemoglobin and hematocrit levels is necessary to manage pregnancy anemia.

The proposed study aims to evaluate healthy lifestyle behaviors, physical activity, and biochemical markers among pregnant women in the first trimester, using various questionnaires and laboratory tests. This study will provide valuable insights into maternal health and guide clinical practices during early pregnancy to reduce complications and enhance overall outcomes.

DETAILED DESCRIPTION:
Pregnancy is a phase in women's lives characterized by psychological, biological, and emotional changes. The process of pregnancy typically spans nine months, divided into three trimesters (Küçükkaya et al., 2018). Identifying risk factors during pregnancy is essential, and these include ethnicity, maternal age, gestational age, antibody presence, iodine sufficiency, parity (number of births), multiple pregnancies, body mass index, and smoking (Curí L.L. et al., 2023). Pregnancy is also linked to various factors that affect a woman's psychological health, family dynamics, and overall quality of life. Pregnant women must collaborate with a multidisciplinary team (doctors, midwives, nurses, physiotherapists, etc.) to manage these risks effectively (Amirshahi et al., 2024).

Pregnant women often experience anxiety about potential negative outcomes during labor and the postpartum period (Küçükkaya et al., 2018). Research indicates that women's concerns and anxieties change across different trimesters (Küçükkaya et al., 2018; Karataylı, S., 2007). Moreover, factors such as age, education level, employment status, and health insurance significantly influence their anxiety levels (Küçükkaya et al., 2018). These concerns-along with anxiety, depression, and stress-affect pregnancy-related responsibilities, nutrition, hygiene, physical activity, travel, and overall acceptance of pregnancy. Therefore, in our study, we plan to assess the healthy lifestyle behaviors of women in their first trimester using the "Pregnancy Healthy Lifestyle Behavior Scale" (Yılmaz E, Karahan N, 2019). This scale, developed by Yılmaz et al., consists of 29 items and 6 subscales (pregnancy responsibility, nutrition, hygiene, physical activity, travel, and pregnancy acceptance) and has undergone validity and reliability testing. It uses a five-point Likert scale, with higher scores indicating more positive health behaviors.

Regular physical activity during pregnancy maintains and improves physical fitness, aids in weight management, reduces the risk of gestational diabetes in obese women, and enhances psychological well-being. It is recommended that women engage in at least 20-30 minutes of moderate-intensity exercise most days of the week. Studies show that physical activity during pregnancy reduces negative outcomes for both the mother and fetus, positively affecting maternal and child health (American College of Obstetricians and Gynecologists, 2015). Physical activity has multiple benefits, including maintaining physical condition, improving quality of life, reducing the risk of obesity-related diseases, and increasing longevity. Generally, physical activity during pregnancy carries minimal risks and benefits most women, particularly those with uncomplicated pregnancies, who are encouraged to engage in personalized exercise programs before, during, and after pregnancy (American College of Obstetricians and Gynecologists, 2015). However, despite its proven benefits, studies have shown that many pregnant women do not engage in adequate physical activity (Göker et al., 2021). Research has found that women's total physical activity levels in the first trimester are lower compared to other trimesters (Lee et al., 2016). Another study shows that physical activity levels increase in the second trimester, with significant improvements noted compared to the first and third trimesters (Özdemir et al., 2017). This decrease in activity in the first trimester may be attributed to efforts to ensure fetal safety and physical discomfort caused by pregnancy (Ko Y-L et al., 2016). However, the pregnancy process is individualized, and some women may engage in regular physical activity even in early pregnancy. Therefore, our study aims to assess physical activity levels in the first trimester. This evaluation will help us understand the frequency of physical activity in early pregnancy and explore its potential effects on pregnancy health. To achieve this, we will use the "Pregnancy Physical Activity Questionnaire" (Chasan-Taber et al., 2004), validated in Turkish by Tosun et al. (2015). This questionnaire consists of 36 items divided into four subscales: occupational activity, household chores, child care, and exercise. The scores will assess the physical activity levels of pregnant women during the first trimester.

Pregnancy also affects thyroid function and can lead to various complications. Factors such as ethnicity, socio-economic status, iodine supplementation, and obesity influence Thyroid-Stimulating Hormone (TSH) levels. Monitoring trimester-specific TSH ranges is important for timely diagnosis and treatment (Yanachkova et al., 2024). Thyroid disorders are common during pregnancy, affecting 2-3% of all pregnancies, with 10% of women having autoimmune thyroid disease despite normal thyroid function. Over the past two decades, a better understanding of thyroid physiology during pregnancy has highlighted the importance of thyroid function adaptation and the negative maternal and neonatal outcomes associated with untreated thyroid disorders, such as hypothyroidism or hyperthyroidism. Increased awareness of thyroid diseases during pregnancy can help reduce complications (Tekin, Y. B., & Güven, E. S. D., 2014). In our study, we will evaluate TSH values during the first trimester.

In addition to thyroid issues, liver dysfunction during pregnancy can be a concern. Around 3% of pregnancies are affected by liver dysfunction (Ch'ng et al., 2002), which can range from mild functional disturbances to rare severe liver diseases. These issues often arise at specific stages of pregnancy. Proper diagnosis and timely treatment are critical for reducing morbidity and mortality risks for both mother and baby (Güven, S., & Türkay, C., 2011). Pregnancy-specific liver diseases can cause changes in liver enzymes such as ALT and AST, which are crucial for identifying complications. Therefore, we will examine ALT and AST levels as part of our study.

Monitoring hemoglobin (HGB) and hematocrit (HCT) levels during pregnancy is crucial for the health of both mother and baby. Low HGB and HCT levels can lead to pregnancy-related anemia. In a study examining multiparous women, the anemia rates based on HGB and ferritin levels were found to be 24.2% and 20.8%, respectively (Çıkım et al., 2020). Higher HGB and HCT levels were found in the control group, while the first trimester group had higher values compared to other trimester groups. In preeclamptic pregnancies, higher levels of HGB and HCT are observed in the umbilical cord (Sürücü et al., 2005).

The required sample size for the study has been calculated using G-power analysis, yielding a total of 649 participants. The study is planned to take place from August 15, 2024, to August 15, 2025, at the Kayseri City Hospital's Obstetrics and Gynecology Clinic and will be a single-center study. Participants will complete the Demographic Information Form, Pregnancy Healthy Lifestyle Behavior Scale, and Pregnancy Physical Activity Questionnaire. Biochemical tests, including complete blood count (CBC) and biochemistry tests, will be performed at the Kayseri City Hospital's Medical Biochemistry Laboratory. CBC results will record HGB and HCT levels, while biochemistry results will record TSH, AST, and ALT levels.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Maternal age between 18 and 40 years
* In the first trimester of pregnancy
* Literate and capable of understanding written materials

Exclusion Criteria:

* Multiple pregnancies
* Non-natural pregnancies
* Family history of thyroid dysfunction
* Presence of thyroid dysfunction and/or autoimmunity
* Clinical diagnosis of Diabetes Mellitus
* Clinical diagnosis of liver disease
* Presence of any physical or mental disability
* Chronic endocrine, autoimmune, or metabolic diseases
* Voluntary withdrawal from the study
* Inability to complete the questionnaires included in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study will be conducted between 15.08.2024 and 15.08.2025. The research will be conducted in Kayseri City Hospital Gynecology and Obstetrics Polyclinic and will be conducted as a single center.
Sampling Method: Non-Probability Sample
Enrollment: 649 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Biochemistry result | 1 day
  LOWER AND UPPER LIMIT VALUES FOR SERUM TSH; 0.1 - 2.5 mU/L for the first trimester, 0.2 - 3.0 mU/L for the second trimester and 0.3 - 3.0 mU/L for the third trimester. Reference values should be between AST: 5-40 U/L and ALT: 7-56 U/L.

SECONDARY OUTCOMES:
Healthy Lifestyle Behaviors Scale During Pregnancy | 1 day (A one-time survey when the patient first arrives)
  "Healthy Lifestyle Behaviors in Pregnant Women Scale" is a five-point Likert-type scale that can be applied to all pregnant women and filled out by the pregnant women themselves. The scale is a measurement tool consisting of a total of 29 items and 6 subscales. Each subscale of the scale can be used alone in studies. Scale items are scored by giving numerical values from 5 to 1 from "always" to "never". There are no reverse-entry items in the scale and high scores obtained from the scale indicate that healthy lifestyle behaviors are positive/high.
Pregnancy Physical Activity Questionnaire | 1 day (A one-time survey when the patient first arrives)
  This scale evaluates 32 activities performed by pregnant women, including housework and care activities, occupational activities, sports and exercise activities, transportation and sedentary life. The intensity of physical activity performed in the scale is expressed as MET (metabolic equivalent). Activity intensities are grouped as sedentary (<1.5 METs), light (1.5-3.0 METs), moderate (3.0-6.0 METs) and vigorous (>0.6 METs).

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kayseri City Hospital, Kayseri, Turkey
  - Kayseri City Hospital, Kayseri